CLINICAL TRIAL: NCT05882942
Title: Effects of Matcha Green Tea on Heart Rate Variability, Substrate Oxidation and Cardiovascular Response at Rest and During Moderate-intensity Exercise in Females
Brief Title: Matcha Green Tea Effects at Rest and During Moderate-intensity Exercise in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chichester (Other)
Responsible Party: Principal Investigator, Mark Eilisabeth Willems, Professor of Exercise Physiology, University of Chichester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 22231905455
Record Dates: First submitted 2023-05-17; First posted 2023-05-31 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: No Condition

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover design
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): Participants will be supplemented with a placebo.
  Interventions: Dietary Supplement: Placebo
- Matcha green tea (Experimental): Participants will be supplemented with Matcha green tea.
  Interventions: Dietary Supplement: Matcha green tea

INTERVENTIONS:
Dietary Supplement: Matcha green tea — This is the condition with the Matcha green tea
  Arms: Matcha green tea
Dietary Supplement: Placebo — This is the condition with the placebo
  Arms: Placebo

SUMMARY:
Intake of the green tea catechin epigallocatechin (EGCG) increased fat oxidation during walking. It is also known to reduce blood pressure and improve body composition. This research will expand the insight on the effects by Matcha green tea supplementation and address the effects on heart rate variability, substrate oxidation at rest, and cardiovascular responses at rest in addition to metabolic and physiologic responses for a 1-hr walk in healthy females.

DETAILED DESCRIPTION:
Intake of the catechin epigallocatechin (EGCG) increased fat oxidation during walking. It is also known to reduce blood pressure and improve body composition. EGCG is the most abundant and potent bioactive compound (50-80% of the total catechin content) found in Matcha green tea (MGT) and is usually consumed as a drink or in a capsulated from unfermented tea leaves. MGT polyphenols have antioxidant and anti-inflammatory properties, providing numerous health benefits, such as the reduced risk of type 2 diabetes and obesity. MGT supplementation (3g over a 24hr period) has been shown to enhance fat oxidation during 30-min brisk walking as well as lower respiratory exchange ratio in females. Understanding the effectiveness of the bioactive compounds found in natural food sources in improving human health is key to informing the general population and the public health policies preceding them; the daily consumption of drinks and food naturally high in EGCG content could be recommended as an essential part of a healthy lifestyle. This research will expand the insight on Matcha green tea supplementation address the effect on heart rate variability, substrate oxidation at rest, and cardiovascular responses at rest in addition to metabolic and physiologic responses for a 1-hr walk in healthy females.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smokers
* not taking any supplements
* no known allergy to green tea

Exclusion Criteria:

* smokers
* known high blood pressure
* on medication

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | Three weeks
  Measurement of root mean square of standard deviation of RR intervals
Carbohydrate oxidation | Three weeks
  Measurement of carbohydrate oxidation in grams/minute
Fat oxidation | Three weeks
  Measurement of fat oxidation in grams/minute
Cardiac output | Three weeks
  Measurement of cardiac output in liters per minute
Stroke volume | Three weeks
  Measurement of stroke volume in milliliters
Total peripheral resistance | Three weeks
  Measurement of total peripheral resistance in (mmHg x min) / mL

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Willems, Principal Investigator — University of Chichester
Locations (2):
- United Kingdom (2):
  - Mark Willems, Chichester, West Sussex
  - University of Chichester, Chichester

IPD SHARING:
Plan to Share IPD: No